CLINICAL TRIAL: NCT04137887
Title: Relative Effectiveness of a High-Dose Quadrivalent Influenza Vaccine Versus a Standard-Dose Quadrivalent Influenza Vaccine in Subjects 65 Years of Age and Older
Brief Title: Study to Evaluate the Effectiveness of a High-Dose Quadrivalent Influenza Vaccine (QIV-HD) Compared to a Standard-Dose Quadrivalent Influenza Vaccine (QIV-SD) in Adults 65 Years of Age and Older
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment terminated due to the COVID-19 pandemic
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QHD00012; 2019-001401-25 (EudraCT Number); U1111-1217-2654 (Other: UTN)
Record Dates: First submitted 2019-10-11; First posted 2019-10-24 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Influenza (Healthy Volunteers)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participants, the outcome assessors in the hospitals and outpatient care, the Investigators, and the Sponsor will remain blinded to the vaccine assignment in order to avoid any bias in reporting and evaluating illnesses or SAEs. An unblinded qualified trial staff member will administer the appropriate vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: QIV-HD (Experimental): Participants received a single injection of 0.7 milliliters (mL) high dose quadrivalent influenza vaccine (QIV-HD), intramuscularly (IM) at Day 0.
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) High-Dose (QIV-HD)
- Group 2: QIV-SD (Active Comparator): Participants received a single injection of 0.5 mL standard-dose quadrivalent influenza vaccine (QIV-SD), IM at Day 0.
  Interventions: Biological: Standard-Dose Inactivated Influenza Vaccine Quadrivalent, Northern Hemisphere strains (QIV-SD)

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) High-Dose (QIV-HD) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular
  Other Names: Efluelda®
  Arms: Group 1: QIV-HD
Biological: Standard-Dose Inactivated Influenza Vaccine Quadrivalent, Northern Hemisphere strains (QIV-SD) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular
  Other Names: VaxigripTetra®
  Arms: Group 2: QIV-SD

SUMMARY:
Primary Objective:

To demonstrate the superior relative effectiveness of QIV-HD as compared to QIV-SD among persons 65 years of age and older for the prevention of cardiovascular and/or respiratory hospitalizations.

Secondary Objective:

* To assess the clinical relative effectiveness of QIV-HD as compared to QIV-SD in prevention of:
* inpatient hospitalization for selected circulatory and respiratory causes
* death, either all-cause or cardiovascular or respiratory causes
* inpatient hospitalization (using primary and secondary discharge diagnoses)
* inpatient hospitalization (using admission diagnoses)
* hospital emergency room visits
* primary care visits to physician or
* major acute cardiovascular events (MACE)
* To assess the characteristics of inpatient hospitalization or hospital emergency room visits or primary care visits to physician by QIV-HD and QIV-SD groups.
* To describe the clinical relative effectiveness of QIV-HD as compared to QIV-SD:
* by age group and by group with specific comorbidities
* for different periods of observation
* To describe all serious adverse events (SAEs) (including adverse event of special interest [AESIs]) for all subjects in both QIV-HD and QIV-SD groups.

DETAILED DESCRIPTION:
Study duration per participant was 1 day of screening and vaccination. The study was planned to be conducted over a period of 3 influenza seasons beginning in 2019-2020. The vaccination period was from October to December.

ELIGIBILITY:
Inclusion criteria:

- Aged 65 years or older on the day of inclusion ("65 years" means from the day of the 65th birthday).

Exclusion criteria:

* Participation at the time of study enrollment (or in the 4 weeks [28 days] preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Previous vaccination against influenza (in the preceding 6 months) with either the study vaccines or another vaccine.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33096 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Investigational Site Number 2469999, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Palmu AA, Pepin S, Syrjanen RK, Mari K, Mallett Moore T, Jokinen J, Nieminen H, Kilpi T, Samson SI, De Bruijn I. High-Dose Quadrivalent Influenza Vaccine for Prevention of Cardiovascular and Respiratory Hospitalizations in Older Adults. Influenza Other Respir Viruses. 2024 Apr;18(4):e13270. doi: 10.1111/irv.13270. PMID 38569647
- [Derived] Hollingsworth R, Palmu A, Pepin S, Dupuy M, Shrestha A, Jokinen J, Syrjanen R, Nealon J, Samson S, De Bruijn I. Effectiveness of the quadrivalent high-dose influenza vaccine for prevention of cardiovascular and respiratory events in people aged 65 years and above: Rationale and design of a real-world pragmatic randomized clinical trial. Am Heart J. 2021 Jul;237:54-61. doi: 10.1016/j.ahj.2021.03.007. Epub 2021 Mar 13. PMID 33722585
- See also: QHD00012 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25340&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at a single site in Finland by Finnish Institute for Health and Welfare in collaboration with multiple health stations overseen by public health care centers in Finland. A total of 33096 participants were enrolled, out of which 1 participant withdrew consent prior to randomization. 33093 participants were vaccinated between 04 November 2019 and 23 December 2019. Among these, 16549 participants were vaccinated in the QIV-HD group and 16544 participants in the QIV-SD group.
Pre-assignment Details: Study was planned to be conducted over a period of 3 influenza seasons beginning in 2019-2020. Enrollment & data collection were disrupted during the 2020-2021 & 2021-2022 influenza seasons due to worldwide coronavirus disease 2019 (COVID-19). Data collection period was chosen as: from 14 days post-vaccination up to end of May of year following vaccination. Study was terminated prematurely after only 1 influenza season (2019-2020) & thus included only season 2019-2020 assessment.
Period: Overall Study
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Started | 16549 | 16546
Vaccinated | 16549 | 16544
Completed | 16445 | 16450
Not Completed | 104 | 96
Not completed — Death | 102 | 92
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all vaccinated participants.
Groups:
- Group 1: QIV-HD: Participants received a single injection of 0.7 mL QIV-HD, IM at Day 0.
- Group 2: QIV-SD: Participants received a single injection of 0.5 mL QIV-SD, IM at Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD | Total
Number analyzed (Participants) | 16549 | 16544 | 33093
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (5.7) | 72.5 (5.6) | 72.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8273 | 8241 | 16514
  Male | 8276 | 8303 | 16579
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospitalizations Due to Cardiovascular or Respiratory Diseases
Description: Number of participants with hospitalizations due to any cardiovascular or respiratory diseases on the basis of International Classification of Diseases, Tenth Revision (ICD-10) codes as per health care professional (HCP) assessment were collected using Finnish health registers and reported in this outcome measure (OM). ICD-10 codes for respiratory system diseases: J00-J06 (acute upper respiratory infections), J09-J18 (influenza & pneumonia), J20-J22 (other acute lower respiratory infections), J40-J47 (chronic lower respiratory diseases), J80-J81 (other respiratory diseases affecting interstitium), J85-J86 (suppurative & necrotic conditions of lower respiratory tract); codes for circulatory diseases: I11 (hypertensive diseases), I20-I25 (ischemic heart diseases), I26-I27 (pulmonary heart disease & diseases of pulmonary circulation), I30, I31, I33, I38-I42, I46-I50 (other forms of heart disease), I63-I67 (cerebrovascular diseases) & I74 (diseases of arteries, arterioles & capillaries).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants | 257 | 272
Statistical Analysis 1: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; Test type: Superiority — Superiority of QIV-HD effectiveness over QIV-SD was demonstrated if the lower bound of the Confidence intervals (CIs) for relative vaccine effectiveness (rVE); expressed in percentage (%) was more than (>) 0%; Relative Vaccine Effectiveness = 5.54, 95% CI 2-sided [-12.43 to 20.66] — rVE: % reduction of 1st occurrence of cardiovascular/respiratory hospitalization cases in QIV-HD group compared to QIV-SD group. 2-sided 95% CIs for rVE was calculated by exact method assuming Binomial distribution of number of cases in both groups

2. Primary Outcome: Number of Participants With Primary Discharge Diagnoses For Any Respiratory and Circulatory Systems Diseases Hospitalizations
Description: Number of participants with primary discharge diagnoses (final diagnosis given to participant before release from hospital) for any respiratory & circulatory diseases hospitalizations on the basis of ICD-10 codes per HCP assessment were collected using Finnish health registers and reported in this OM. ICD-10 codes for respiratory system diseases were: J00-J06 (acute upper respiratory infections), J09-J18 (influenza & pneumonia), J20-J22 (other acute lower respiratory infections), J40-J47 (chronic lower respiratory diseases), J80-J81 (respiratory diseases affecting interstitium), J85-J86 (suppurative & necrotic conditions of the lower respiratory tract); and codes for circulatory system diseases were: I11 (hypertensive diseases), I20-I25 (ischemic heart diseases), I26-I27 (pulmonary heart disease & diseases of pulmonary circulation), I30, I31, I33, I38-I42, I46-I50 (other heart disease), I63-I67 (cerebrovascular diseases) and I74 (diseases of arteries, arterioles and capillaries).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Any diseases of the respiratory system | 88 | 93
  Any diseases of the circulatory system | 171 | 184
Statistical Analysis 1: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; Statistical analysis for diseases of respiratory system; Test type: Superiority — Superiority of QIV-HD effectiveness over QIV-SD was demonstrated if the lower bound of the CIs for rVE, expressed in % was > 0%; Relative Vaccine Effectiveness = 5.40, 95% CI 2-sided [-27.99 to 30.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1: QIV-HD vs Group 2: QIV-SD; Statistical analysis for diseases of circulatory system; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Relative Vaccine Effectiveness = 7.09, 95% CI 2-sided [-15.04 to 25.00] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Primary Discharge Diagnoses for Various Respiratory and Circulatory Diseases
Description: Number of participants with primary discharge diagnoses (final diagnosis given to participant before release from hospital) due to each disease of respiratory and circulatory system on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM. The codes selected were pneumonia (J12-J18); heart failure (I50); acute myocardial infarction (I21); atrial fibrillation and flutter (I48); cerebral infarction (I63); influenza and pneumonia (J09-J18) and influenza (J09-J11).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Pneumonia | 62 | 62
  Heart failure | 27 | 27
  Acute myocardial infarction | 31 | 40
  Atrial fibrillation and flutter | 40 | 32
  Cerebral infarction | 27 | 28
  Influenza and pneumonia | 62 | 62
  Influenza | 6 | 8

4. Secondary Outcome: Number of Participants With Deaths
Description: Number of participants reporting death (all-cause) and due to any diseases of respiratory and circulatory system and separately due to each disease on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM. Based on ICD-10 codes, codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85-J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. Codes for pneumonia (J12-J18); heart failure (I50); acute myocardial infarction (I21); atrial fibrillation and flutter (I48); cerebral infarction (I63); influenza and pneumonia (J09-J18) and influenza (J09-J11).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Death (All-cause) | 102 | 92
  Death due to any diseases of respiratory system | 3 | 9
  Death due to any diseases of circulatory system | 19 | 16
  Death due to Pneumonia | 3 | 9
  Death due to Heart failure | 3 | 1
  Death due to Acute myocardial infarction | 0 | 4
  Death due to Atrial fibrillation and flutter | 0 | 0
  Death due to Cerebral infarction | 1 | 1
  Death due to Influenza and pneumonia | 3 | 9
  Death due to Influenza | 0 | 0

5. Secondary Outcome: Number of Participants With Primary and Secondary Admission Diagnoses for Respiratory and Circulatory Diseases
Description: Number of participants with primary admission diagnosis (diagnosis given to the participant at the time of admission to hospital) and secondary admission diagnosis (diagnosis that coexist with the primary admission diagnosis at the time of admission) due to any diseases of respiratory and circulatory system and separately for each disease on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM. ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. Codes for pneumonia (J12-J18); heart failure (I50); acute myocardial infarction (I21); atrial fibrillation and flutter (I48); cerebral infarction (I63); influenza and pneumonia (J09-J18) and influenza (J09-J11).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Any diseases of the respiratory system | 102 | 110
  Any diseases of the circulatory system | 195 | 199
  Pneumonia | 69 | 72
  Heart failure | 45 | 43
  Acute myocardial infarction | 27 | 37
  Atrial fibrillation and flutter | 60 | 51
  Cerebral infarction | 22 | 34
  Influenza and pneumonia | 69 | 72
  Influenza | 7 | 7

6. Secondary Outcome: Number of Participants With Primary and Secondary Discharge Diagnoses for Respiratory and Circulatory Diseases
Description: Number of participants with primary discharge diagnosis (final diagnosis given to a participant before release from the hospital) and secondary discharge diagnosis (diagnoses that coexist with the primary discharge diagnosis at the time of discharge) due to any diseases of respiratory and circulatory system and separately for each disease on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM. ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. Codes for pneumonia (J12-J18); heart failure (I50); acute myocardial infarction (I21); atrial fibrillation and flutter (I48); cerebral infarction (I63); influenza and pneumonia (J09-J18) and influenza (J09-J11).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Any diseases of the respiratory system | 130 | 143
  Any diseases of the circulatory system | 257 | 263
  Pneumonia | 72 | 78
  Heart failure | 46 | 57
  Acute myocardial infarction | 38 | 41
  Atrial fibrillation and flutter | 105 | 99
  Cerebral infarction | 29 | 34
  Influenza and pneumonia | 72 | 78
  Influenza | 9 | 9

7. Secondary Outcome: Number of Participants With Hospital Emergency Room Visits
Description: Number of participants reporting hospital emergency room visits due to any diseases of respiratory and circulatory system and separately due to each disease, on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM. ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. Codes for pneumonia (J12-J18); heart failure (I50); acute myocardial infarction (I21); atrial fibrillation and flutter (I48); cerebral infarction (I63); influenza and pneumonia (J09-J18) and influenza (J09-J11).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Any diseases of the respiratory system | 95 | 97
  Any diseases of the circulatory system | 158 | 158
  Pneumonia | 28 | 36
  Heart failure | 15 | 11
  Acute myocardial infarction | 0 | 0
  Atrial fibrillation and flutter | 109 | 118
  Cerebral infarction | 1 | 0
  Influenza and pneumonia | 28 | 36
  Influenza | 5 | 10

8. Secondary Outcome: Number of Participants With Acute Primary Care Visits to Physician
Description: Number of participants reporting acute primary care visits to physician due to any diseases of the respiratory and circulatory system and separately for each disease, on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM. ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. Codes for pneumonia (J12-J18); heart failure (I50); acute myocardial infarction (I21); atrial fibrillation and flutter (I48); cerebral infarction (I63); influenza and pneumonia (J09-J18) and influenza (J09-J11).
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Any diseases of the respiratory system | 279 | 285
  Any diseases of the circulatory system | 137 | 120
  Pneumonia | 23 | 25
  Heart failure | 16 | 19
  Acute myocardial infarction | 3 | 5
  Atrial fibrillation and flutter | 63 | 53
  Cerebral infarction | 2 | 2
  Influenza and pneumonia | 23 | 25
  Influenza | 3 | 1

9. Secondary Outcome: Number of Participants With Major Acute Cardiovascular Events (MACE)
Description: Major acute cardiovascular events (MACE) were defined by all of the following outcomes: ischemic heart diseases based on codes I20-I25, non-fatal myocardial infarction based on codes I21-I23, unstable angina based on codes I20 and I25 and fatal or non-fatal cerebral infarction based on code I63. Number of participants with MACE events on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and reported in this OM.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Ischaemic heart diseases | 46 | 68
  Myocardial infarction | 31 | 40
  Unstable angina | 16 | 30
  Cerebral infarction | 27 | 28

10. Secondary Outcome: Percentage of Observed Cardiorespiratory Events During the Assessment Period
Description: Percentage of observed cardiorespiratory events during the different time durations over the assessment period were reported in this OM. The following codes were taken into account: ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. International Classification of Primary Care Second Edition (ICPC-2) codes: R72, R74 to R81, R83, R95 and R96; K70, K74 to K80, K82, K84, K87 and K90 to K93.
Time Frame: 14 to 30 days, 31 to 60 days, 61 to 90 days, 91 to 120 days and 121 days or above
Population: Analysis was performed on all vaccinated participants.
Measure: Number; unit: percentage of events
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
percentage of events
  14 to 30 days | 11.83 | 10.20
  31 to 60 days | 18.93 | 19.44
  61 to 90 days | 17.20 | 20.49
  91 to 120 days | 19.93 | 18.65
  121 days or above | 32.12 | 31.22

11. Secondary Outcome: Duration of Cardiorespiratory Hospitalization
Description: Duration (in days) of cardiorespiratory hospitalization was defined as stop date of event (hospitalization) minus start date of event plus 1. The following codes were taken into account: ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants. Here 'overall number of participants analyzed'= participants with available data for this OM.
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 257 | 272
days | 5.0 [2 to 84] | 5.0 [2 to 60]

12. Secondary Outcome: Number of Participants With Hospitalizations Due to Cardiovascular or Respiratory Diseases: By Age Groups
Description: Number of participants with hospitalizations due to any diseases of the respiratory or circulatory system and separately for respiratory and circulatory diseases on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and presented by age groups (65 to 74 years, 75 years and above and 85 years and above) in this OM. The following codes were taken into account: ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  65 to 74 years: Any diseases of respiratory/circulatory system | 120 | 151
  65 to 74 years: Diseases of respiratory system | 42 | 48
  65 to 74 years: Diseases of circulatory system | 78 | 105
  75 years and above: Any diseases of respiratory/circulatory system | 137 | 121
  75 years and above: Diseases of respiratory system | 46 | 45
  75 years and above: Diseases of circulatory system | 93 | 79
  85 years and above: Any diseases of respiratory/circulatory system | 32 | 32
  85 years and above: Diseases of respiratory system | 6 | 15
  85 years and above: Diseases of circulatory system | 26 | 18

13. Secondary Outcome: Number of Participants With Hospitalizations Due to Cardiovascular or Respiratory Diseases: Groups With Specific Comorbidities
Description: Number of participants with hospitalizations due to any diseases of the respiratory or circulatory system and separately for respiratory and circulatory diseases on the basis of ICD-10 codes as per HCP assessment were collected using Finnish health registers and presented by various comorbidities (diabetes, cardiovascular history and chronic lung disease) in this OM. The following codes were taken into account: ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85 and J86; and codes for any circulatory system diseases were: I11, I20-I25, I26, I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  Any diseases of respiratory/circulatory system with comorbidity diabetes | 60 | 63
  Diseases of circulatory system with comorbidity diabetes | 34 | 44
  Diseases of respiratory system with comorbidity diabetes | 26 | 21
  Any diseases of respiratory/circulatory system with comorbidity of chronic lung disease | 54 | 57
  Diseases of circulatory system with comorbidity of chronic lung disease | 26 | 21
  Diseases of respiratory system with comorbidity of chronic lung disease | 28 | 37
  Any diseases of respiratory/circulatory system with comorbidity of cardiovascular history | 104 | 108
  Diseases of circulatory system with comorbidity of cardiovascular history | 77 | 82
  Diseases of respiratory system with comorbidity of cardiovascular history | 27 | 28

14. Secondary Outcome: Number of Occurrences for Cardiorespiratory Diseases During Influenza Epidemic Period
Description: The influenza epidemic period as per Finnish epidemic thresholds was defined as the period where the influenza incidence was high. The following codes were taken into account: ICD-10 codes for any respiratory system diseases were: J00-J06, J09-J18, J20-J22, J40-J47, J80-J81, J85-J86; and codes for any circulatory system diseases were: I11 and I16, I20-I25, I26-I27, I30, I31, I33, I38-I42, I46-I50, I63-I67 and I74. ICPC-2 codes: R72, R74 to R81, R83, R95 and R96; K70, K74 to K80, K82, K84, K87 and K90 to K93.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Data for this outcome measure was not collected and analyzed as influenza epidemic period was not observed before study termination.
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Serious Adverse Reactions (SARs), and Adverse Event of Special Interest (AESIs)
Description: SAE: any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization/ prolongation of existing hospitalization, resulted in persistent/ significant disability/ incapacity, was congenital anomaly/ birth defect or was an important medical event. SAR: all noxious and unintended responses to study vaccine related to any dose administered that resulted in death, was life-threatening, required hospitalization/ prolongation of existing hospitalization, resulted in persistent/ significant disability/ incapacity, or was congenital anomaly or birth defect. SAR referred to potential causal relationship between study vaccine & SAE, based on assessment of healthcare professional. AESI was defined as one of scientific & medical concern specific to study for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was considered appropriate. Relatedness to study vaccine was based on Investigator's discretion.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants
  SAE | 109 | 98
  AESI | 4 | 6
  SAR | 1 | 1

16. Secondary Outcome: Number of Participants With Non-fatal SAEs
Description: SAEs were defined as any untoward medical occurrence that at any dose was life-threatening, required inpatient hospitalization/ prolongation of existing hospitalization, resulted in persistent/ significant disability/ incapacity, was congenital anomaly/ birth defect or was an important medical event. Information on non-fatal SAEs was collected from the health registers.
Time Frame: From 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD | Group 2: QIV-SD
Number analyzed (Participants) | 16549 | 16544
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Reported adverse events data was collected from 14 days post-vaccination up to 31 May 2020 post-vaccination (i.e., up to a duration of 6 months post-vaccination)
Description: Analysis was performed on all vaccinated participants.
Groups:
- Group1: QIV-HD: Participants received a single injection of 0.7 mL QIV-HD, IM at Day 0.
Arm/Group | Group1: QIV-HD | Group 2: QIV-SD
All-Cause Mortality (participants affected / at risk) | 102/16549 | 92/16544
Serious Adverse Events (participants affected / at risk) | 109/16549 | 98/16544
Other Adverse Events (participants affected / at risk) | 0/16549 | 0/16544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1: QIV-HD (N=16549) | Group 2: QIV-SD (N=16544)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 4 (4) | 2 (2)
Congestive Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 13 (13) | 2 (2)
Hypertensive Heart Disease (Cardiac disorders) | 2 (2) | 2 (2)
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 3 (3)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 2 (2) | 2 (2)
Sudden Cardiac Death (General disorders) | 0 (0) | 1 (1)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 9 (9)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure To Extreme Temperature (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Appendix Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bronchioloalveolar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gingival Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haematopoietic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant Neoplasm Of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Neoplasm Papilla Of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Respiratory Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral T-Cell Lymphoma Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Bell's Palsy (Nervous system disorders) | 3 (3) | 6 (6)
Cerebral Haemorrhage (Nervous system disorders) | 5 (5) | 3 (3)
Cerebral Infarction (Nervous system disorders) | 3 (3) | 0 (0)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertensive Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Physical Assault (Social circumstances) | 0 (0) | 1 (1)
Aortic Aneurysm Rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic Dissection Rupture (Vascular disorders) | 0 (0) | 2 (2)
Aortic Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
COVID-19 severely impacted the study resulting in low influenza circulation and disruption of trial recruitment for subsequent seasons (no enrollment done for seasons 2020-21 & 2021-22). Moreover, the events collected as primary outcomes could have been driven by COVID cases, diluting the effect of influenza vaccines on such events. The study was prematurely terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT04137887/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT04137887/SAP_001.pdf